CLINICAL TRIAL: NCT05267704
Title: Evaluating the Feasibility of Virtual Reality for Procedural Sedation in Pediatric Renal Biopsy Patients
Brief Title: Evaluating the Feasibility of VR for Pediatric Renal Biopsies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-35095
Record Dates: First submitted 2021-10-07; First posted 2022-03-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Pain, Procedural; Procedural Anxiety; Sedation Complication
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- VR Arm (Experimental): Pediatric patients age 5-17 using the VR headset during renal biopsy.
  Interventions: Device: Samsung Gear Virtual Reality Headset

INTERVENTIONS:
Device: Samsung Gear Virtual Reality Headset — VR headset displaying preselected game during renal biopsy

SUMMARY:
The purpose of this study is to assess the use of virtual reality (VR) as an adjunct or alternative to pharmacologic sedation in pediatric patients undergoing renal biopsy.

DETAILED DESCRIPTION:
Children aged 5-17 scheduled for renal biopsy will be offered the option to use a virtual reality (VR) headset that displays an interactive game as part of their renal biopsy experience. The standard of care of sedation medications will still be available to patients who are unable to complete the procedure with only the VR headset without pharmacologic sedation. Pain and anxiety will be monitored continuously using validated scales by a pediatric hospitalist and sedation nurse. These providers, as well as patients and parents, may ask for additional medications for adequate analgesia and anxiolysis.

ELIGIBILITY:
Inclusion Criteria:

- Patients age 5-17 receiving a renal biopsy at the University of California, San Francisco (UCSF) Benioff Children's Hospital

Exclusion Criteria:

* Patients who cannot lie supine for their renal biopsy will be excluded from the study
* Patients with injuries to the head/face that would prohibit wearing a headset
* Patients with loss of consciousness, altered mental status, life-threatening injuries/illness or multi-trauma
* Patients with open skin, lice, scabies, or other infectious skin conditions on the head/face
* Patients with a history of or current symptoms of vertigo
* Patients who are blind
* Patients with significant developmental or cognitive delays who may not be able to engage with or tolerate the virtual reality environment, as determined by their parent/caregiver
* Patients on whom the VR headset does not fit appropriately

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of VR to Patients/Families | From arrival to procedural room to completion of procedure (~30 minutes)
  Acceptability of VR as non-pharmacologic sedation based on a team-made Likert scale survey given to patients, parents, and providers (Likert scale, with 1 = "strongly disagree" as most dissatisfied with VR experience and 5 = "strongly agree" as most satisfied with VR experience and a better perceived outcome

SECONDARY OUTCOMES:
Pre- and Post-Procedural Pain (Change in Observation Scale of Behavioral Distress Scale) | From arrival to procedural room to completion of procedure (~30 minutes), at 15-second intervals
  Pain as recorded on Observation Scale of Behavioral Distress (OSBD 11 point behavioral scale rating the number and intensity of distress behaviors demonstrated before/during/after the procedure in 15-second intervals; higher scores and intensity of distress behaviors indicate worse pain)
Pre- and Post-Procedural Anxiety (Change in Childhood Anxiety Meter) | From arrival to procedural room to completion of procedure (~30 minutes)
  Anxiety as recorded on Childhood Anxiety Meter (CAM 0-10 scale, using analogy of mercury thermometer to ask children to rate level of anxiety, with higher score indicating more anxiety)
Pre- and Post-Procedural Anxiety (Change in Child Fear Scale) | From arrival to procedural room to completion of procedure (~30 minutes)
  Children's Fear Scale (CFS 0-4 scale, visual face scale correlated with 0-4 numeric scale, with 4 being highest fear/anxiety related to procedure)
Patient, Parent, and Provider Satisfaction (Post-procedure) | From arrival to procedural room to completion of procedure (~30 minutes)
  Patient, parent, and provider satisfaction as assessed on 4-question Likert scale (0 to 5, with 5 being high satisfaction) survey
Total Dose of Sedation Needed | From arrival to procedural room to completion of procedure (~30 minutes)
  Total dose (mg/kg) of pharmacologic sedation needed to complete renal biopsy with adequate patient analgesia, anxiolysis, and comfort

CONTACTS AND LOCATIONS:
Overall Officials: Justin Libaw, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Benioff Children's Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jung MJ, Libaw JS, Ma K, Whitlock EL, Feiner JR, Sinskey JL. Pediatric Distraction on Induction of Anesthesia With Virtual Reality and Perioperative Anxiolysis: A Randomized Controlled Trial. Anesth Analg. 2021 Mar 1;132(3):798-806. doi: 10.1213/ANE.0000000000005004. PMID 32618627
- [Background] Taylor JS, Chandler JM, Menendez M, Diyaolu M, Austin JR, Gibson ML, Portelli KI, Caruso TJ, Rodriguez S, Chao SD. Small surgeries, big smiles: using virtual reality to reduce the need for sedation or general anesthesia during minor surgical procedures. Pediatr Surg Int. 2021 Oct;37(10):1437-1445. doi: 10.1007/s00383-021-04955-6. Epub 2021 Jul 16. PMID 34269867
- [Background] Goldman RD, Behboudi A. Virtual reality for intravenous placement in the emergency department-a randomized controlled trial. Eur J Pediatr. 2021 Mar;180(3):725-731. doi: 10.1007/s00431-020-03771-9. Epub 2020 Aug 10. PMID 32779029
- See also: Samsung Gear VR Headset — https://www.samsung.com/global/galaxy/gear-vr/